CLINICAL TRIAL: NCT03675828
Title: Virtual Visits in Heart Failure Care Transitions
Acronym: VIV-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wilson Tang, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-651
Record Dates: First submitted 2018-08-27; First posted 2018-09-18 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Heart Failure
Keywords: Heart Failure; Distance Health; Virtual Health
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Visit (Experimental): In this arm, the 7-day post discharge visit will be completed by a scheduled virtual visit with a member of the study team using the Cleveland Clinic Online Express Care application on a computer or a tablet/phone.
  Interventions: Behavioral: Virtual Visit
- Outpatient Clinic (No Intervention): In this arm, the 7-day post discharge visit will be completed by a standard-of-care, in-person outpatient visit with a member of the study team in the heart failure clinic.

INTERVENTIONS:
Behavioral: Virtual Visit — The Cleveland Clinic Express Care Online application will be used in this intervention. The subjects will have a virtual consult with a clinician from the study team that will mirror an experience had at an outpatient post-discharge visit, including review of systems and medications.
  Arms: Virtual Visit

SUMMARY:
This study evaluates the use of virtual visits in the post-discharge care of patients with heart failure. Participants admitted to the hospital with a primary diagnosis of heart failure will be randomized at discharge to either a virtual visit or outpatient visit for their 7-day post discharge follow up visit.

DETAILED DESCRIPTION:
Published guidelines recommend that patients being discharged home after hospitalization for HF should be offered a 7-day post-discharge outpatient clinic visit as a way to increase engagement with care and reduce risk of poor outcomes. Unfortunately no-show rates for the 7-day post-discharge outpatient visit in this population are high, suggesting poor engagement. The investigators have previously observed a 76% no-show rate at the Cleveland Clinic Main Campus. This study is to evaluate whether use of 7-day post-discharge virtual visit versus in-person visit can improve adherence with post-discharge appointment.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized for primary diagnosis of HF;
2. Anticipated to be discharged home;
3. Agreeable to longitudinal post-discharge care at Cleveland Clinic Main Campus in the first few weeks after hospital discharge;
4. Patient or an individual in their social support network has the ability (equipment and connectivity) to do a virtual visit after hospital discharge;

Exclusion Criteria:

1. Being transferred to another hospital, or being discharged to an inpatient facility or nursing home;
2. Being discharged to hospice;
3. Subject currently enrolled in an interventional research study that requires an in-person clinical visit within 7 days post-discharge.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Proportion of completed post discharge visits via virtual visit or in outpatient setting | 12 months
  Proportion of patients who complete 7-day post discharge appointment (virtually or in-person)

SECONDARY OUTCOMES:
45-day unplanned readmission and death measures stratified by visit method (virtually or in-person) | 12 months
  Composite and individual components of unscheduled all-cause first occurrence of (a.) hospital readmission, (b.) emergency department visit, or (c.) death, in the first 45 days after hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Hong Wilson Tang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorodeski EZ, Moennich LA, Riaz H, Jehi L, Young JB, Tang WHW. Virtual Versus In-Person Visits and Appointment No-Show Rates in Heart Failure Care Transitions. Circ Heart Fail. 2020 Aug;13(8):e007119. doi: 10.1161/CIRCHEARTFAILURE.120.007119. Epub 2020 Jul 30. No abstract available. PMID 32762457